CLINICAL TRIAL: NCT04800731
Title: Study of Lymphopenia as a Specific Biomarker or Prognostic Risk Factor for Disease Severity in Elderly Patients With COVID-19.
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Nathalie compté, Clinic head of geriatric unit, Universitair Ziekenhuis Brussel
Other Study IDs: Lymfopenia
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Lymphopenia; Covid19; Older People
Keywords: lymphopenia; Covid 19; Older People
MeSH Terms: conditions — Lymphopenia; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Group 1 will consist of 100 patients COVID-19 positive patients older than 70 years old hospitalized in UZ Brussel from February 2020 until September 2020 with a positive RT-PCR test for SARS-CoV-2.
  Interventions: Other: observation no intervention
- Group 2: Group 2 will consist of 100 patients older than 70 years old hospitalized in UZ Brussel for acute infections other than COVID-19.
  Interventions: Other: observation no intervention
- Group 3: Group 3 will consist of healthy aged people defined as in the modified SENIEUR protocol (12, 13). This group is recruited from a previously conducted study. These are community dwelling individuals above the age of 70 and considered as almost healthy with some conditions that are present in the majority of old people such as osteoporosis, osteoarthritis or atherosclerosis.
  Interventions: Other: observation no intervention

INTERVENTIONS:
Other: observation no intervention — no intervention

SUMMARY:
Background: Lymphopenia is reported to be associated with the severity of disease progression in COVID-19. Low lymphocyte count is also associated with increasing age. No study has yet investigated the effects of lymphopenia in this disease on the outcome in elderly people.

Objectives: To assess the outcome of lymphopenia in elderly patients having COVID-19 and its usefulness as prognostic factor in elderly people.

Methods: Retrospective cohort study. Clinical data (medical history, comorbidities, treatments, geriatric syndromes) and biological parameters will be collected from 100 hospitalized geriatric COVID-19 patients (> 70 yrs.) (Group 1) and 100 hospitalized geriatric patients (> 70 yrs.) presenting with acute infection other than COVID-19 (Group 2) and will be compared according to the presence/absence of lymphopenia. A third Group (3) will be studied to assess the influence of comorbidities on lymphopenia consisting of healthy aged elderly (> 70 yrs.).

DETAILED DESCRIPTION:
Introduction In December 2019 a cluster of viral pneumonia cases in Wuhan, a city in the Hubei Province of China, led to the discovery of a novel pathogen that was later named Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) (1). SARS-CoV-2 rapidly spread throughout the population of China and subsequently to all continents of the world (except for Antarctica). On 11 March 2020 the outbreak was declared a pandemic by the World Health Organisation (WHO) (2). In September confirmed cases have been reported from 217 different countries and has resulted in over 27 million infected individuals and as near as 900.000 deadly cases reported to the WHO (3, 4). SARS-CoV-2 does not discriminate between social status, age or ethnicity and an effective treatment remains absent until so far. However, risk factors associated with severity of disease progression have been identified and include advanced age (>65y), comorbidities with inclusion of arterial hypertension, cardiovascular disease, cerebrovascular disease, respiratory disease and laboratory parameters such as low CD3+CD8+ T cells (<75 cells.µL-1), low lymphocyte count, neutrophil to lymphocyte ratio (N/L) (N/L ratio >3.13) and increased cardiac troponin I (≥0.05ng.mL-1) (5-9).

It has been demonstrated that both age and lymphopenia are risk factors associated with severity of disease progression in COVID-19 patients. A low lymphocyte count, however, is also known to be associated with increasing age in healthy individuals (10). Another study has also shown that a high CRP was associated with lymphopenia in a geriatric hospitalized population before the apparition of COVID-19 (11). This observation raises the question whether or not lymphopenia is a specific prognostic marker for the COVID-19 illness in elderly patients.

The aims of this study are:

1. to assess the specificity of lymphopenia in COVID-19 cases in elderly people thanks to the comparison of 3 Groups:

   1. Group 1 consists of COVID-19 cases
   2. Group 2 consists of patients with an acute infection other than COVID-19
   3. Group 3 consists of healthy aged people defined as in the modified SENIEUR protocol
2. to assess the correlation of lymphopenia in COVID-19 cases and the outcome
3. to assess the relationship between other morbidities (such as CV diseases / risk factors) and lymphopenia in elderly people.

Patients and methods

Patients:

To assess the outcome of lymphopenia in COVID-19 infections in elderly patients, three Groups will be studied:

Group 1 will consist of 100 patients COVID-19 positive patients older than 70 years old hospitalized in UZ Brussel from February 2020 until September 2020 with a positive RT-PCR test for SARS-CoV-2.

Group 2 will consist of 100 patients older than 70 years old hospitalized in UZ Brussel for acute infections other than COVID-19. To avoid including false negative patients, these patients will be selected from January 2019 until December 2019, before the first COVID-19 cases were documented in Belgium. An acute infection other than COVID-19 will be defined as 1) viral infection confirmed by nasopharynx swab for: influenza, RSV, parainfluenza, rhinoviruses, coronaviruses or 2) bacterial infection confirmed with positive blood culture, positive articular punction, positive expectorations, pneumonia on chest radiograph, or infection documented by abdominal imagery (CT or echo), a positive urine culture with a confirmed pyelonephritis with a renal echography or a DMSA scintigraphy or specific clinical symptoms for pyelonephritis and positive hemoculture. A positive urine culture alone is not considered as urine infection because of the high prevalence of asymptomatic bacteriuria in geriatric patients.

To assess the influence of comorbidities on lymphopenia in elderly people, the Groups 1 and 2 will be compared to a well-defined historical group (Group 3):

Group 3 will consist of healthy aged people defined as in the modified SENIEUR protocol (12, 13). This group is recruited from a previously conducted study. These are community dwelling individuals above the age of 70 and considered as almost healthy with some conditions that are present in the majority of old people such as osteoporosis, osteoarthritis or atherosclerosis.

Inclusion criteria Cfr definition of the three groups Exclusion criteria Patients receiving immunosuppressive therapy, patients with known active cancer or hematologic disorders, patients undergoing radio- or chemotherapy or with known autoimmune diseases will not be included since these underlying conditions or therapies can interfere with white blood cell count in a way that is beyond the scope of this research.

Methods:

Determination of clinical characteristics All subjects will be assessed for underlying illnesses by medical archives and blood sampling. Social evaluation included determination of age, gender and home (private versus institution). Clinical data included smoking and alcohol habits, body mass index (BMI), medical history, current treatment and reasons for hospitalization. Cardiovascular (CV) diseases are defined as a history of stroke, myocardial infarct, cardiac insufficiency (assessed by anterior cardiac echography and clinical symptoms), cerebral vascular disease or atheromatosis assessed by carotid or leg Doppler ultrasonography and ischemic symptoms. CV risk factors will be defined by the presence in the medical history of arterial hypertension (AHT), type 2 diabetes mellitus (DM 2), hypercholesterolemia or statin intake, infarct history or smoking.

Comprehensive geriatric assessment When possible, we will obtain a comprehensive geriatric assessment: The comorbidities and the severity of the medical problems were scored using the "Cumulative Illness Rating Scale-Geriatric" (CIRS-G), which is an instrument to quantify disease burden. It differentiates older adults with the highest risk and severity of infection with a markedly impaired vaccine response (14). It comprises a comprehensive review of medical problems of 14 organ systems. It is based on a 0 to 4 rating of each organ system (15). The "Geriatric Depression Scale" was used to assess the risk of depression (GDS-15) in 15 questions (16). The assessment of "Activities of Daily Living" (ADL) was made using Katz's scale. It includes the following items: bathing, dressing, transfer, toilet, continence and eating. Each task is graded on a 4-level scale (1 to 4 for Katz's scale), where lower levels represent the absence of dependence and upper levels the maximal dependence for the task (17). Cognitive functions were assessed using the "Mini Mental State Examination" (MMSE). Possible scores range from 0 to 30 points, with scores<24/30 indicating impaired cognitive function (18). Nutritional status was assessed using the "Malnutrition Universal Screening Tool" (MUST) (19). Social complexity was defined by the need for an intervention with a social worker (need for home care, rehabilitation nursing home or financial help). The sum of geriatric syndrome includes the following: fall, social complexity, delirium, undernutrition, dependence, depression, dysphagia, incontinence, orthostatic hypotension, inappropriate prescription, and cognitive dysfunction.

Biological parameters Data from the routine biochemical assessment performed in the first 24 hrs and after 3 to 5 days after admission to a geriatric unit will be collected (total and differential white blood cell counts, hemoglobin and hematocrit, renal function and electrolytes CRP, albumin, prealbumin, vitamin B12, and folic acid levels).

Outcome:

To assess the outcome of patients with or without lymphopenia, the number of rehospitalisation's, the admissions to an intensive care unit, the complications such as lung embolism, the duration of the hospital stay, the mortality, the place of the discharge and the severity score of the CT scan of the thorax in COVID-19 + patients will be collected.

Procedures This is a retrospective study. No interventions will be performed.

Flowchart

Study analysis Statistical analysis IBM SPSS version 25 will be used for statistical analyses. The Kolmogorov-Smirnov test will be used to determine the normality of the data.

Mann Whitney rank sum test for non-parametric data or a student T-test for parametric data will be performed to compare patients with and without lymphopenia for COVID-19, other infections, comorbidities, complications, geriatric assessment, duration of hospitalisation, rehospitalisation, mortality, place of discharge.

In order to identify clinical and biological factors that could be significantly associated with lymphopenia, we performed univariate analyses (depicted by Pearson's coefficient). For all volunteers, these parameters comprised CV diseases and risk factors (smoking, arterial hypertension, type 2 diabetes, cholesterol levels, BMI), COVID-19, other infections, comorbidities, complications, geriatric assessment, duration of hospitalisation, rehospitalisation, mortality, place of discharge.

In order to define independent predictive factors of lymphopenia, we tested several models by stepwise backward multi-linear regression analyses.

ELIGIBILITY:
Inclusion Criteria:

Cfr definition of the three groups

Exclusion Criteria:

* Patients receiving immunosuppressive therapy, patients with known active cancer or hematologic disorders, patients undergoing radio- or chemotherapy or with known autoimmune diseases will not be included since these underlying conditions or therapies can interfere with white blood cell count in a way that is beyond the scope of this research.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Group 1 will consist of 100 patients COVID-19 positive patients older than 70 years old hospitalized in UZ Brussel from February 2020 until September 2020 with a positive RT-PCR test for SARS-CoV-2.
  Group 2 will consist of 100 patients older than 70 years old hospitalized in UZ Brussel for acute infections other than COVID-19.
  To assess the influence of comorbidities on lymphopenia in elderly people, the Groups 1 and 2 will be compared to a well-defined historical group (Group 3):
  Group 3 will consist of healthy aged people defined as in the modified SENIEUR protocol (12, 13). This group is recruited from a previously conducted study. These are community dwelling individuals above the age of 70 and considered as almost healthy with some conditions that are present in the majority of old people such as osteoporosis, osteoarthritis or atherosclerosis.
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
assess the specificity of lymphopenia in COVID-19 cases in elderly people | 3 years
  to assess the specificity of lymphopenia in COVID-19 cases in elderly people, thanks to the comparison of 3 Groups:
  1. Group 1 consists of COVID-19 cases
  2. Group 2 consists of patients with an acute infection other than COVID-19
  3. Group 3 consists of healthy aged people defined as in the modified SENIEUR protocol

SECONDARY OUTCOMES:
to assess the correlation of lymphopenia in COVID-19 cases and the outcome | 3 years
  2) to assess the correlation of lymphopenia in COVID-19 cases and the outcome, we will compare the group number 1 with the group number 2
to assess the relationship between other morbidities (such as CV diseases / risk factors) and lymphopenia in elderly people. | 3 years
  to assess the specificity of lymphopenia in COVID-19 cases in elderly people, thanks to the comparison of 3 Groups:
  1. Group 1 consists of COVID-19 cases
  2. Group 2 consists of patients with an acute infection other than COVID-19
  3. Group 3 consists of healthy aged people defined as in the modified SENIEUR protocol

CONTACTS AND LOCATIONS:
Locations (1):
- UZ brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
There is no sharing plan